CLINICAL TRIAL: NCT02050139
Title: A PROSPECTIVE, RANDOMIZED, DOUBLE-BLIND, CROSS-OVER STUDY TO EVALUATE THE RENAL AND BIOHUMORAL EFFECTS OF L-CYSTEINE COMPARED TO PLACEBO IN STABLE PERITONEAL DIALYSIS PATIENTS WITH RESIDUAL DIURESIS
Brief Title: L-Cysteine in Peritoneal Dialysis
Acronym: CINDY
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mario Negri Institute for Pharmacological Research (Other)
Collaborators: Bio3 Research s.r.l. - Milan Italy (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Supportive Care
Other Study IDs: CINDY
Record Dates: First submitted 2014-01-28; First posted 2014-01-30 (Estimated); Last update posted 2015-06-30 (Estimated); Status verified 2015-06

CONDITIONS: Uremia
Keywords: L-Cysteine; Peritoneal dialysis; Diuresis; Glomerular filtration rate; Peritoneal function; Inflammation
MeSH Terms: conditions — Uremia; Inflammation | interventions — Cysteine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- L-cysteine (Biocysan®) (Experimental): Study subjects will take one tablet of L-cysteine or placebo every morning four times a week and two tablets of L-cysteine or placebo three times a week during the whole study period
  Interventions: Dietary Supplement: L-cysteine
- Placebo (Placebo Comparator): Study subjects will take one tablet of L-cysteine or placebo every morning four times a week and two tablets of L-cysteine or placebo three times a week during the whole study period
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: L-cysteine
  Other Names: Biocysan®
  Arms: L-cysteine (Biocysan®)
Other: Placebo
  Arms: Placebo

SUMMARY:
Over the last decades, peritoneal dialysis has grown worldwide to become one of the most common modalities of renal replacement therapy, particularly in developing or newly industrialized countries, such as India, China, Korea, Turkey, Malaysia, Mexico and Brazil. Peritoneal dialysis has been associated with an initial survival benefit compared to hemodialysis, although this advantage becomes less apparent over time, likely due to the progressive loss of residual renal function and the development of pathological alterations of peritoneum . Recent results suggest that an antioxidant therapy by N-acetyl-cysteine oral supplementation may improve residual renal function in peritoneal dialysis patients. This finding may have major clinical relevance, as preserving residual renal function in peritoneal dialysis patients has been associated with improved survival . Aim of the present randomized, double-blind, crossover study is to confirm the preliminary evidence of the beneficial effects of antioxidant agents on residual renal function by using the L-enantiomeric form of cysteine in 10 prevalent peritoneal dialysis patients with residual diuresis.

ELIGIBILITY:
Inclusion Criteria:

* Males and females aged ≥ 18 years;
* Chronic automated peritoneal dialysis;
* Residual 24-hour diuresis ≥ 100 ml with less than 30% changes over the three months preceding randomization;
* Written informed consent.

Exclusion Criteria:

* Chronic automated peritoneal dialysis therapy since less than three months;
* Diabetes mellitus;
* Acute peritonitis during the three months before enrollment;
* Concomitant treatment with other antioxidant agents (including N-acetyl-cysteine and vitamin C);
* Cystinuria;
* Pregnancy or breastfeeding;
* Childbearing potential without reliable contraceptive methods during the whole study period;
* Alcohol or drug (excluding tobacco) abuse;
* Inability to comply with the study procedures during the whole study period, legal incapacity;
* Cancer and any severe systemic disease or clinical condition that may jeopardize data interpretation or completion of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2014-02; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
24-hour urine output | Changes from Baseline at 1,2 and 3 month.
Measured Glomerular Filtration Rate (GFR) | Changes from baseline at 1, 2 and 3 month.

SECONDARY OUTCOMES:
Office systolic, diastolic, pulse and mean blood pressure | Changes from Baseline at 1,2 and 3 month.
Urinary albumin excretion. | Changes from Baseline at 1,2 and 3 month.
2.27% Peritoneal Equilibration test (PET) | Changes from Baseline at 1,2 and 3 month.
Pulse wave velocity (measured by tonometry) | Changes from Baseline at 1,2 and 3 month.
Augmentation Index (measured by tonometry) | Changes from Baseline at 1,2 and 3 month.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Research Center for Rare Diseases, Ranica, Bergamo, Italy